CLINICAL TRIAL: NCT01867736
Title: BIOTRONIK's - First in Men Study of the Passeo-18 LUX Drug Releasing PTA Balloon Catheter vs. the Uncoated Passeo 18 Balloon Catheter in Subjects Requiring Revascularization of Infrapopliteal Arteries (BIOLUX P-II).
Brief Title: BIOLUX P-II First-in-Man Study to Compare the Passeo-18 Lux DRB Against POBA in Infrapopliteal Arteries
Acronym: BIOLUX P-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C1102
Record Dates: First submitted 2013-05-27; First posted 2013-06-04 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Atherosclerosis; Arteriosclerosis; Vascular Disease; Peripheral Artery Disease
Keywords: Stenosis; Occlusions; Infrapopliteal arteries; Below the knee arteries; PTA; POBA; DRB
MeSH Terms: conditions — Atherosclerosis; Arteriosclerosis; Vascular Diseases; Peripheral Arterial Disease; Constriction, Pathologic; Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Passeo-18 Lux DRB (Experimental): Passeo-18 Lux Drug Releasing Balloon catheter
  Interventions: Device: Passeo-18 Lux DRB
- Standard PTA (POBA) (Active Comparator): Uncoated Passeo-18 PTA balloon catheter
  Interventions: Device: Standard PTA (POBA)

INTERVENTIONS:
Device: Passeo-18 Lux DRB
  Other Names: Passeo-18 LUX Drug Releasing PTA Balloon Catheter
  Arms: Passeo-18 Lux DRB
Device: Standard PTA (POBA)
  Other Names: Uncoated Passeo-18 PTA balloon catheter
  Arms: Standard PTA (POBA)

SUMMARY:
A prospective, multicentric, randomized controlled trial to assess the safety and performance of the Passeo-18 Lux Paclitaxel releasing PTA balloon catheter versus the uncoated Passeo 18 PTA balloon catheter for the treatment of stenosis, restenosis or occlusion of the infrapopliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent.
2. Subject is willing and able to comply with follow-up evaluations.
3. Subject is ≥ 18 years old.
4. Single or sequential de novo or restenotic lesions (stenosis ≥ 70% diameter reduction or occlusion) in the infrapopliteal arteries ≥ 30 mm. Lesions should not extend beyond the ankle joint.
5. A maximum of 2 different vessels can be treated: successful wire crossing is required for the first target vessel before randomization occurs.
6. Subject with PAD or critical limb ischemia according to the current guidelines in need for urgent revascularization to relieve symptoms and improve walking capacity.
7. Reference Vessel Diameter (RVD) 2 - 4 mm, based on visual estimation.
8. Inflow free from flow-limiting lesion confirmed by angiography. Patients with flow-limiting inflow lesions (> 50% stenosis) can be included if lesion(s) have been treated successfully before the index procedure, with a maximum residual stenosis of 30% per visual assessment.
9. At least one non-occluded crural vessel with angiographically documented run-off to the foot.
10. Successful wire crossing of the lesion.

Exclusion Criteria:

1. Flow-limiting (> 50% DS) inflow lesion proximal to target lesion, left untreated.
2. Failure to obtain <30% residual stenosis in a pre-existing haemodynamically significant (>50% DS) inflow lesion (DEB or DES not allowed for the treatment of inflow lesions).
3. Infrapopliteal lesions extending beyond the ankle joint and involving crural vessels.
4. Acute thrombus in the target vessel (eg complication of inflow lesion treatment) documented by angiogram, if not treated successfully prior to enrolment).
5. Planned major amputation above the ankle of target limb, or any other planned major surgery within 30 days post-procedure.
6. Previous bypass surgery of target vessel.
7. Previously implanted stent in target lesion.
8. Haemorrhagic diathesis or coagulopathy or other disorders such as gastrointestinal ulcerations or cerebral disorders that would restrict prescription of dual anti-platelet therapy.
9. Subject with hepatic failure, deep vein thrombosis, thrombophlebitis, systemic lupus erythematous or subject is on immunosuppressant therapy.
10. Subject with acute MI ≤ 3 months.
11. Renal failure with a creatinine of ≥ 2,5 mg/dl, except patients currently on regular dialysis.
12. Phenprocoumon intake, except for patients who are treated for Arterial Fibrillation. For these patients Phenprocoumon treatment can be interrupted and re-started after treatment with Dual Antiplatelet Therapy for 4 weeks post procedure.
13. Known allergy to contrast media used for angiography that cannot be controlled by pre-medication with steroids and/or antihistaminica.
14. Allergy, intolerance or hypersensitivity to Paclitaxel or related compounds and/or to the delivery matrix n-Butyryl tri-n-hexyl citrate(BTHC).
15. Co- morbid conditions limiting life expectancy ≤ 1 year.
16. Patients that are under active treatment for cancer; Patients, who have been successfully treated for cancer in the past, can be included.
17. Subject is participating in another clinical device trial where the primary endpoint has not yet been reached.
18. Pregnant and/or breast-feeding females or females who intend to become pregnant during the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-07; Primary Completion 2014-01 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Safety: Major adverse event rate (MAE), defined as all cause death, major amputation of target extremity, target lesion thrombosis, target lesion revascularisation (TLR)and target vessel revascularization (TVR) at 30 days. | 30 days
Performance: Target lesion primary patency rate at 6 months assessed by quantitative vascular angiogram (QVA). | 6 months

SECONDARY OUTCOMES:
Target lesion failure, assessed by target lesion revascularization (TLR) rate at 6 months and 12 months | 6 and 12 months
Target vessel revascularization (TVR) rate at 6 months and 12 months | 6 and 12 months
Binary re-stenosis rate at 6 months, assessed by QVA | 6 months
Major adverse event rate, defined as all cause death, major amputation of target extremity, target lesion thrombosis, TLR and TVR at 6 months and 12 months | 6 and 12 months
Change in mean ABI at discharge, 30 days, 6 months and 12 months | Discharge, 30 days, 6 months and 12 months
Change in Rutherford classification at 30 days, 6 months and 12 months | 30 days, 6 months and 12 months
Quality of life evaluation, assessed by EQ5D questionnaire at baseline, 30 days, 6 months and 12 months | Baseline, 30 days, 6 months and 12 months
Duplex based primary patency at 30 days, 6 months and 12 months | 30 days, 6 months and 12 months
Procedural success, defined as successful vascular access, completion of endovascular procedure and immediate morphologic success with a residual stenosis <30%. | Day 0
Device success, defined as exact deployment according to Instructions For Use | Day 0
Technical success, defined as device or procedural success without the occurrence of major adverse events during the hospital stay. | Participants will be followed for the duration of hospital stay, an expected average of 1-2 days
Late Lumen Loss | 6-months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Universitäts-Herzzentrum Freiburg - Bad Krozingen, Germany
Locations (6):
- Medical University of Graz, Graz, Austria
- Belgium (2):
  - Imelda Hospital, Bonheiden
  - A.Z. Sint-Blasius, Dendermonde
- Germany (3):
  - Universitäts-Herzzentrum Freiburg, Bad Krozingen
  - Gefaesszentrum Berlin, Medizinische Klinik, Ev. Krankenhaus Königin Elisabeth Herzberge, Berlin
  - Parkkrankenhaus Leipzig Südost GmbH, Leipzig